CLINICAL TRIAL: NCT05491616
Title: Nivolumab During Active Surveillance After Neoadjuvant Chemoradiation for Esophageal Cancer: SANO-3 Study
Acronym: SANO-3
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. B. (Bianca) Mostert, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-6KC
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer
Keywords: immunotherapy; Nivolumab
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Nivolumab; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab q4w (Experimental): patients will receive Nivolumab at 480mg Q4W starting 10-14 weeks
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — In this SANO-3 study, patients will receive Nivolumab at 480mg Q4W starting 10-14 weeks after nCRT (i.e., when cCR has been established) until disease progression or unacceptable toxicity, for a maximum duration of 1 year.
  Other Names: Immune Checkpoint Inhibitor

SUMMARY:
In an effort to prevent surgery in selected patients with esophageal cancer, the SANO-2 study offers active surveillance to patients with clinically complete response (cCR) after neoadjuvant chemoradiation (nCRT). Some of these patients will never develop locoregional and/or distant recurrence of disease (persistent cCR). However, two-thirds of the patients that undergo active surveillance still get disease recurrence. This can be locoregional regrowth or distant metastases. To increase the efficacy of active surveillance (reduce the proportion of patients that need surgery) and improve survival, effective systemic maintenance therapy is needed. The CheckMate 577 randomized, placebo controlled, clinical trial showed that Nivolumab increases disease free survival in patients after nCRT and esophagectomy.

Objective: To assess the efficacy of nivolumab during active surveillance in patients with cCR after neoadjuvant chemoradiation for esophageal cancer

DETAILED DESCRIPTION:
The rationale of maintenance nivolumab in patients with cCR undergoing active surveillance is to decrease the risk for disease recurrence and improve survival as well as to optimize the chance for having an organ sparing treatment. In this non-randomized phase II study we will assess the efficacy of maintenance nivolumab in patients who are undergoing active surveillance after nCRT in the context of the SANO-2 trial: the SANO-3 study. The SANO-3 study aims to identify a new indication for immunotherapy in primary esophageal cancer: patients who have been identified as a clinical complete responders 10-14 weeks after nCRT can be included. This subgroup of patients will not undergo standard surgery but instead continue with active surveillance after nCRT when they opt for participation in the SANO-2 trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Written informed consent and ability to understand the nature of the study and the study-related procedures and to comply with them
3. Histologically proven, resectable adenocarcinoma or squamous cell carcinoma of the esophagus or GEJ (gastroesophageal junction) according to the UICC TNM7 definition. Tumors of the esophagus and tumors of which the epicentre is within 5 cm of the GEJ are eligible for inclusion in the trial (Type 1 and Type 2 according to Siewert classification of esophagogastric adenocarcinoma
4. Pre-treatment stage cT2-4aN0-2M0 disease. In case of stage cT4a, the possibility for a curative resection has to be explicitly verified by the multidisciplinary tumor board
5. nCRT (CROSS regimen) completed, i.e. all radiotherapy fractions administered.
6. Complete clinical response 10-14 weeks after nCRT as determined by endoscopy with biopsies, EUS with FNA and PET/CT scanning
7. No prior cytotoxic chemotherapy other than as part of the neoadjuvant chemoradiation (CROSS)
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
9. Adequate cardiac function (cardiac function tests such as echocardiography only necessary in symptomatic patients).
10. Adequate respiratory function (pulmonary function tests only necessary in symptomatic patients).
11. Adequate bone marrow function (White Blood Cells >2x10^9/l; Haemoglobin >6,2mmol/L; platelets >100x10^9/l). In the event of transfusions, the last red blood cell transfusion should be more than 2 weeks before inclusion.
12. Adequate renal function (Glomerular Filtration Rate >40 ml/min) or Serum creatinine <=1.5 x upper limit of normal (ULN)
13. Adequate liver function (AST and ALT < 3.0 x ULN; Total bilirubin < 1.5 x ULN (except participants with Gilbert Syndrome who may have a total bilirubin level of < 3.0 x ULN)
14. Women of child-bearing potential must have a negative serum pregnancy test during screening period
15. Patients must be willing to use adequate contraception during the study and for 3 months after the end of the study.

Exclusion Criteria:

1. Language difficulty, dementia or altered mental status prohibiting the understanding and giving of informed consent and to complete quality of life questionnaires;
2. Patients who were treated with definitive chemoradiotherapy
3. Patients who were unable to complete all radiotherapy fractions of the nCRT
4. No cCR at 10-14 weeks
5. Esophageal cancer evaluated as not curatively-resectable by the multidisciplinary tumour board, for instance because ingrowth in the trachea, aorta or vertebra (cT4b)
6. Gastric carcinoma
7. Clinically significant (active) cardiac disease (e.g. symptomatic coronary artery disease or myocardial infarction within last 12 months)
8. Clinically significant lung disease (Forced Expiratory Volume in one second (FEV1)
9. Pregnant and lactating women, or patients of reproductive potential who are not using effective birth control methods. If barrier contraceptives are used, they must be continued by both sexes throughout the study.
10. Participation, current or during the last 30 days prior to informed consent, in another intervention trial with interference to the chemotherapeutic or chemoradiotherapeutic intervention of this study.
11. Expected lack of compliance with the protocol
12. Refusal to undergo further active surveillance (i.e., opting for esophageal resection)
13. Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured or successfully resected, such as basal or squamous cell skin cancer, superficial bladder cancer, or GC, or carcinoma in situ of the prostate, cervix, or breast
14. Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
15. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents for adults, or > 0.25 mg/kg daily prednisone equivalent for adolescent) or other immunosuppressive medications within 14 days of study treatment. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents for adults, or > 0.25 mg/kg daily prednisone equivalent for adolescents are permitted, in the absence of active autoimmune disease.
16. Participants who received prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
17. Anti-tumor treatment other than as part of neoadjuvant chemoradiation (CROSS) within 28 days of first administration of study treatment
18. Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
19. Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g, hepatitis B surface antigen (HBsAg, Australia antigen) positive, or hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative)
20. Participants must not have received a live / attenuated vaccine within 30 days of first treatment.
21. History of severe hypersensitivity reactions to other monoclonal antibodies
22. History of allergy or hypersensitivity to study drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Disease Free survival 18 months | 18 months
  No locoregional or distant recurrence of disease, evaluated by PETCT, EUS (Endoscopic Ultrasound), endoscopy + bite-on-bite biopsy

SECONDARY OUTCOMES:
the proportion of patients with locoregional and/or distant metastase | occurence or end of follow-up (2 years after start immunotherapy), which comes first
  Locoregional or distant recurrence of disease, evaluated by PETCT, EUS (Endoscopic Ultrasound), endoscopy + bite-on-bite biopsy
the proportion of patients that undergo esophagectomy | occurence or end of follow-up (2 years after start immunotherapy), which comes first
  For locoregional disease recurrence, evaluated at pre-specified time points
health-related quality of life (HRQOL) at baseline, 3, 6, 12 and 24 months after inclusion | baseline, 3, 6, 12 and 24 months after inclusion
  The EORTC QLQ-C30 questionnaire will be used. Scale scores will be calculated following the scoring guidelines of the EORTC questionnaires. Scores will be summarized by means of the appropriate descriptive statistics (mean + SD or median + IQR) at each measurement point.
overall survival at 2 years | 2 years
  No recurrence of disease at 2 years, evaluated by PETCT, EUS (Endoscopic Ultrasound), endoscopy + bite-on-bite biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Mostert, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands